CLINICAL TRIAL: NCT01887769
Title: Body Composition Analysis for Patient With Lung Cancer Using Computed Tomography Image Analysis
Acronym: BAT-SCAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Didier Saey, PhD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Other Study IDs: 20824
Record Dates: First submitted 2013-02-13; First posted 2013-06-27 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Body composition analysis; Ct-Scan; Muscle mass; Cachexia
MeSH Terms: conditions — Lung Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung cancer patient at diagnosis

SUMMARY:
Rationale: With 1.6 million new cases diagnosed each year and 1.3 million deaths, lung cancer is the leading cancer-related death worldwide and it represents a pressing health issue. Patients with lung cancer are more likely to experience cachexia, a severe debilitating disorder causing fatigue, weight loss, muscle wasting and associated with reduced physical function, increased chemotherapy toxicity and reduced survival. This syndrome occurring in about 80% of advanced cancer patients is the direct cause of death in about 20% of cases. However, despite the importance of cachexia in lung cancer, it has been mainly studied from several assessment methods which do not usually differentiate muscle from other tissues.

Aim: To analyze body composition of patients with lung cancer at diagnosis using computed tomography (CT-Scan) image analysis.

Methods: This is a retrospective study extending over a period of 3 years conducted at the Institut universitaire de cardiologie et de pneumologie de Québec (2009-2012). We listed patients newly diagnosed with lung cancer who had a thoraco-abdominal CT-scan performed in our institution. Following the collection of clinical data from patient records, we used SliceOmatic software to quantify muscle area, visceral fat area and subcutaneous fat area from a single abdominal cross-sectional image at the level of the third lumbar vertebra.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Between 40-80 years of age
* Primary lung cancer diagnosed between 2009 and 2012
* CT-Scan done at the time of the diagnosis

Exclusion Criteria:

* Chemotherapy, radiotherapy or surgery at the time of the first Ct-Scan image
* History of other cancer (during the last five years)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients, at diagnosis, following in oncology clinic
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change of muscle area (cm2/m2) at the level of the third lumbar vertebra | at the time of the diagnosis of lung cancer and one year following it.
Change of fat area (cm2/m2) at the level of the third lumbar vertebra | at the time of the diagnosis of lung cancer and one year following it.

SECONDARY OUTCOMES:
days of survival | From the time of the diagnosis of lung cancer until one year

CONTACTS AND LOCATIONS:
Overall Officials: Didier Saey, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada